CLINICAL TRIAL: NCT04044937
Title: Fluoroethyltyrosine for the Evaluation of Intracranial Neoplasm
Brief Title: Fluoroethyltyrosine for Evaluation of Intracranial Neoplasms
Acronym: UC-GlioFET
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Hope (Other)
Responsible Party: Sponsor-Investigator, Thomas Hope, Assistant Professor, University of California, San Francisco
Organization: University of California, San Francisco (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 171022; NCI-2018-01875 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2019-07-25; First posted 2019-08-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Intracranial Neoplasm; Low Grade Glioma; Recurrent Glioblastoma; Recurrent World Health Organization (WHO) Grade II Glioma; Recurrent WHO Grade III Glioma
MeSH Terms: conditions — Brain Neoplasms; Glioblastoma | interventions — (18F)fluoroethyltyrosine; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Population 1: Intracranial neoplasms (glial or metastatic disease) (Experimental): Participants with intracranial neoplasms (glial or metastatic disease) with concern for recurrence or progression on conventional imaging (e.g., MRI) will receive F-18 fluoroethyltyrosine (FET) injected intravenously over approximately 1 minute and receive a single PET image lasting up to 40 minutes. Repeat FET PET will be offered to adult patients.
  Interventions: Drug: F-18 Fluoroethyltyrosine (FET); Procedure: Positron Emission Tomography (PET)
- Population 2: Suspected glial neoplasms (Experimental): Participants with suspected glial neoplasms (Grade 2-4) planning to undergo a non-investigational biopsy or surgery prior to non-investigational, primary treatment (radiation therapy and/or surgery) will receive F-18 fluoroethyltyrosine (FET) injected intravenously over approximately 1 minute and receive a single PET image lasting up to 40 minutes. Repeat FET PET will be offered to adult patients.
  Interventions: Drug: F-18 Fluoroethyltyrosine (FET); Procedure: Positron Emission Tomography (PET)

INTERVENTIONS:
Drug: F-18 Fluoroethyltyrosine (FET) — Patients given an injected dose of 4 to 7 millicurie (mCi) of FET per scan. The radiopharmaceutical will be administered while the patient is in the PET scanner
  Other Names: 18F-FET; 18FET; 2''-[F18] Fluoro-ethyl-L-tyrosine; [18F]-Fluoro-ethyl-L-tyrosine; Fluorine-18 2''-Fluoroethyl-L-tyrosine; Fluoroethyltyrosine F18; O-(2[F18]fluoroethyl)-L-tyrosine
Procedure: Positron Emission Tomography (PET) — All patients receive single PET imaging lasting for 40 minutes. Acquired PET data will be reconstructed so that three time points are created: (1) Perfusion: 60-second acquisition that starts immediately when activity is noted in the field of view, (2) Equilibrium: 10-minute acquisition acquired between 10 and 20 minutes after injection, and (3) Washout: 10-minute acquisition acquired between 30 and 40 minutes after injection. A repeat PET image will be offered to adult patients.
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron Emission Tomography; Positron Emission Tomography Scan; proton magnetic resonance spectroscopic imaging

SUMMARY:
This phase II trial studies how well F-18 fluoroethyltyrosine (fluoroethyltyrosine) works in detecting tumors in participants with intracranial tumors that have come back. FET accumulates in malignant cells within intracranial neoplasms and can be used to detect recurrent disease and characterize the grade of glial neoplasms. Imaging agents such as FET can help oncologist to see the tumor better during a positron emission tomography (PET) scan.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if F-18 fluoroethyltyrosine (FET) PET can differentiate between benign treatment-related changes and recurrence in comparison to pathology in population 1 with recurrent metastatic disease and high-grade gliomas.

II. To determine if FET PET can accurately differentiate between low-grade and high-grade gliomas in population 2.

SECONDARY OBJECTIVES:

I. To determine if FET PET can differentiate between benign treatment-related changes and recurrence in comparison to pathology or imaging follow-up in population 1.

II. To determine if FET PET can differentiate between benign treatment-related changes and recurrence in comparison to pathology in population 1 with recurrent low-grade gliomas.

OUTLINE:

Participants receive F-18 fluoroethyltyrosine intravenously (IV) over approximately 1 minute and undergo PET over 40 minutes. After completion of study treatment, participants are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Age > 3 years.
* Presence or suspicion of intracranial neoplasm in two populations.

  * Population 1: Patients after primary treatment (radiation therapy and/or surgery) with suspicion of recurrence on magnetic resonance imaging (MRI). Three sub-populations will be considered:

    * Recurrent metastatic lesions.
    * Recurrent high-grade gliomas (grades 3 and 4).
    * Recurrent low-grade gliomas (grades 1 and 2).
  * Population 2: Patients prior to primary treatment with planned biopsy or surgical resection.

Exclusion Criteria:

* Patient with known incompatibility to PET or computed tomography (CT)/MRI scans.
* Patient unlikely to comply with study procedures, restrictions and requirements and judged by the investigator to be unsuitable for study participation.

  * Sedation or anesthesia can be used for patients who cannot tolerate the exam.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-03-31 (Actual)

PRIMARY OUTCOMES:
Misclassification rate for either having recurrent disease or not having recurrent disease for patients previously treated for glial and metastatic disease (Population 1) | Up to 6 months
  Radiologists will classify lesions as having recurrent disease or not having recurrent disease. True Positives (TP) are defined as an FET PET read positive for tumor and pathology/follow-up demonstrates tumor recurrence in at least one biopsy sample, False positives (FP) are defined as an FET PET read positive for tumor and pathology/follow-up demonstrates negative tumor recurrence in all of the biopsy samples, True negatives (TN) are defined as an FET PET read as negative for tumor and pathology/follow-up also negative tumor recurrence in all of the biopsy samples and a false negative (FN) is defined as an FET PET read as negative for tumor and pathology/follow-up demonstrates tumor recurrence in at least one biopsy sample. Misclassification rate = [FP+FN)]/[FP+FN+TP+TN]
Misclassification rate for either high grade or low grade in patients with suspected neoplasms (Population 2) | Up to 6 months
  Readers will have access only to FET PET images for participants with suspected glial neoplasms (Grade 2-4) planning to undergo biopsy or surgery prior to primary treatment during evaluation and will grade the lesions in a binary fashion as having Grade II glial neoplasms or having Grade III/IV glial neoplasms. True positive (TP2): FET PET read as positive for Grade III/IV neoplasm, pathology demonstrates Grade III/IV neoplasm. False positive (FP2): FET PET read as positive for Grade III/IV neoplasm, pathology demonstrates Grade II neoplasm. True negative (TN2): FET PET read as positive for Grade II neoplasm, pathology demonstrates Grade II neoplasm. False negative (FN2): FET PET read as positive for Grade II neoplasm, pathology demonstrates Grade III/IV neoplasm. Misclassification rate = [FP2+FN2]/[FP2+FN2+TP2+TN2]

SECONDARY OUTCOMES:
Binary characterization of follow-up imaging as positive/negative for tumor recurrence | Up to 6 months
  Participants with available histology (performed within 4 weeks of FET scans) or follow-up imaging (performed within 6 months of FET scan) will be included and a composite truth standard for recurrence or treatment-related changes will be evaluated for each case. In the absence of pathology, the composite truth standard will use available clinical information to make a determination. Positive for tumor recurrence on follow-up imaging will be based on Response assessment in neuro-oncology criteria (RANO) criteria reads. Follow-up imaging has to be performed within six months of the FET PET imaging study to be considered for evaluation. Additionally, the composite truth standard may consider tumor board notes and subsequent management of the patient to make a determination.
Misclassification rate for FET PET in the evaluation of recurrent low-grade gliomas (Population 1) | Up to 6 months
  Low-grade glioma is defined by low uptake of FET. Radiologists will classify lesions based on imaging as either having recurrent disease or not having recurrent disease. True Positives (TP1L) are defined as an FET PET read positive for low-grade tumor and pathology/follow-up demonstrates low-grade tumor recurrence in at least one biopsy sample, False positives (FP1L) are defined as an FET PET read positive for low grade tumor recurrence and pathology/follow-up demonstrates negative low-grade tumor recurrence in all of the biopsy samples, True negatives (TN1L) are defined as an FET PET read as negative for low-grade tumor recurrence and pathology/follow-up also negative for low grade tumor recurrence in all of the biopsy samples and a false negative (FN1L) is defined as an FET PET read as negative for low grade tumor recurrence and pathology/follow-up demonstrates low grade tumor recurrence in at least one biopsy sample. Misclassification rate = [FP1L+FN1L)]/[FP1L+FN1L+TP1L+TN1L]
Degree of inter-rater reliability for tracer uptake | Up to 6 months
  Fleiss' kappa statistic will be used to determine the agreement between the assessment of FET-PET tumor targeting (tracer uptake in target lesion: yes/ no), as assessed by three independent blinded readers. Scores range from 0 to 1 with higher scores indicating a great degree of agreement
Degree of inter-rater reliability for radiological interpretations | Up to 6 months
  Cohen's kappa statistics will be used to determine the reproducibility of the assessment by individual readers when analyzing the same data repeatedly and measures the agreement between two raters who each classify items into mutually exclusive categories.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Hope, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-21): https://cdn.clinicaltrials.gov/large-docs/37/NCT04044937/Prot_SAP_000.pdf